CLINICAL TRIAL: NCT06009211
Title: Impact of Aromatherapy on Nausea in Hospitalized Children Undergoing Rehabilitation: A Nurse-led Approach
Brief Title: Impact of Aromatherapy on Nausea in Hospitalized Children Undergoing Rehabilitation
Status: Enrolling by invitation | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, AustinLovenstein, Submitted on behalf of Laikin Ulrich, RN IV Care Coordinator, Acute Care Rehabilitation, Arkansas Children's Hospital Research Institute
Other Study IDs: 275439
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Nausea
Keywords: kids; nausea; aromatherapy; rehabilitation
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aromatherapy: Randomized crossover research study
  Interventions: Other: QueaseEase

INTERVENTIONS:
Other: QueaseEase — Study participants will participate in one week with aromatherapy treatment and one week without aromatherapy treatment (randomly ordered) to serve as their own control.

SUMMARY:
Children, ages 8 - 17, will be enrolled in a research study about the impact of aromatherapy on nausea in the pediatric rehabilitation unit.

DETAILED DESCRIPTION:
Children will participate in the study for two weeks. One week the child will receive a aromatherapy product for nausea and the other week the child will not receive the product.

If this aromatherapy is effective at decreasing nausea, the child may be more likely to participate in their rehabilitation therapy sessions. Information gathered during the study may potentially benefit other patients by helping to develop hospital practices of using aromatherapy in the pediatric rehabilitation unit.

Children participating in the study may or may not help the child but may help children in the future:

1. Children may have less nausea, which could help them feel better, more likely to participate in their rehabilitation activities, and may be able to take better care of themselves.
2. Children may have a reduction in the need for taking medications that help nausea.
3. The research may benefit children in the future by helping to develop hospital practices about using aromatherapy in pediatric rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 8 to 17 years of age on the rehabilitation unit and service at Arkansas Children's Hospital
* Patients with a Glascow Coma Scale (GCS) of 13-15
* Patients with a Rancho Los Amigos Revised Scale score of 5 or higher
* Ability to read and write in English
* Patient to have an expected length of stay of at least 2 weeks

Exclusion Criteria:

* Patients with any mechanical or obstructive pathophysiology (appendicitis, bowel obstruction, or intussusception, etc.)
* Known allergy or sensitivity to lavender, peppermint, spearmint, or ginger
* Patients with known asthma and/or pulmonary conditions
* Wards of the State or any other agency or institution

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted on a 10 bed pediatric rehabilitation unit at Arkansas Children's Hospital. The goals of inpatient rehabilitation are to assist patients in reaching their greatest level of independence and to maximize each child's recovery. Admission criteria include: 1) a medically stable patient who is able and willing to actively participate in 3 hours of therapy (combined time for occupational, physical and speech therapy) per day, 6 days a week; 2) a diagnosis where the patient is expected to benefit from a comprehensive inpatient interdisciplinary rehabilitation program; and, 3) established goals that are specific and pertain to improving functional independence. The top three diagnoses for children admitted to the rehabilitation unit include ABI, TBI, and spinal cord injury. Other diagnoses include, but are not limited to, amputation, burn injury, and cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Wellbeing | Two week duration
  Is there an improvement in overall wellbeing as evidenced by a rate of change in nausea with the implementation of aromatherapy in pediatric patients on an inpatient rehabilitation unit?
  The Baxter Animated Retching Faces (BARF) scale will be used along with a patient diary where patients record how they are feeling. The BARF scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).

SECONDARY OUTCOMES:
Symptoms of Nausea | Two week duration
  To measure the impact of aromatherapy on the overall wellbeing, specifically the symptoms associated with nausea, of pediatric patients on the inpatient rehabilitation unit measured by the Baxter Animated Retching Faces (BARF) scale as compared to standard therapy.
  The Baxter Animated Retching Faces (BARF) scale will be used along with a patient diary where patients record how they are feeling. The BARF scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).
Change in Nausea | Two week duration
  To measure the impact of aromatherapy on the overall wellbeing as evidenced by a rate of change in nausea of pediatric patients on the inpatient rehabilitation unit measured by the frequency of antiemetic medication administration as compared to standard therapy.
  The Baxter Animated Retching Faces (BARF) scale will be used along with a patient diary where patients record how they are feeling. The BARF scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).

CONTACTS AND LOCATIONS:
Overall Officials: Laikin Ulrich, BSN, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arruda J, Yeh AM. Integrative Approach to Pediatric Nausea. Pediatr Ann. 2019 Jun 1;48(6):e236-e242. doi: 10.3928/19382359-20190517-01. PMID 31185115
- [Background] Baxter AL, Watcha MF, Baxter WV, Leong T, Wyatt MM. Development and validation of a pictorial nausea rating scale for children. Pediatrics. 2011 Jun;127(6):e1542-9. doi: 10.1542/peds.2010-1410. Epub 2011 May 29. PMID 21624874
- [Background] Brown L, Danda L, Fahey TJ 3rd. A Quality Improvement Project to Determine the Effect of Aromatherapy on Postoperative Nausea and Vomiting in a Short-Stay Surgical Population. AORN J. 2018 Oct;108(4):361-369. doi: 10.1002/aorn.12366. PMID 30265393
- [Background] Czarnecki ML, Michlig JR, Norton AM, Stelter AJ, Hainsworth KR. Use of Aromatherapy for Pediatric Surgical Patients. Pain Manag Nurs. 2022 Dec;23(6):703-710. doi: 10.1016/j.pmn.2022.08.003. Epub 2022 Sep 16. PMID 36123297
- [Background] Marsh E, Millette D, Wolfe A. Complementary Intervention in Postoperative Care: Aromatherapy's Role in Decreasing Postoperative Nausea and Vomiting. J Holist Nurs. 2022 Dec;40(4):351-358. doi: 10.1177/08980101211065555. Epub 2021 Dec 15. PMID 34905993
- [Background] Sanchez FA, Rosales JR, Godoy PR, Barria RM. Effects of inhalation aromatherapy as a complementary therapy in pediatric patients in the clinical practice: A systematic review. Complement Ther Clin Pract. 2022 Feb;46:101516. doi: 10.1016/j.ctcp.2021.101516. Epub 2021 Nov 23. PMID 34837806
- [Background] Weaver MS, Robinson J, Wichman C. Aromatherapy improves nausea, pain, and mood for patients receiving pediatric palliative care symptom-based consults: A pilot design trial. Palliat Support Care. 2020 Apr;18(2):158-163. doi: 10.1017/S1478951519000555. PMID 31423959